CLINICAL TRIAL: NCT01999296
Title: Prospective Evaluation of the Use of Thunderbeat Vessel Sealing Device in Laparoscopic Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cantonal Hosptal, Baselland (Other)
Responsible Party: Principal Investigator, Daniel Steinemann, MD, Principal Investigator, Cantonal Hosptal, Baselland
Other Study IDs: Thunderbeat in Laparoscopy
Record Dates: First submitted 2013-11-15; First posted 2013-12-03 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Indication for Laparoscopic Surgery (Any)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing laparoscopic surgery
  Interventions: Device: Use of Thunderbeat (TM) in laparoscopic surgery

INTERVENTIONS:
Device: Use of Thunderbeat (TM) in laparoscopic surgery

SUMMARY:
All patients undergoing laparoscopic visceral and gynecologic procedures using the combined bipolar and ultrasonic vessel sealing and dissection device Thunderbeat are entered in a prospective registry. Data will be analysed concerning the safe use of the instrument and perioperative blood loss.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing laparoscopic visceral or gynecologic surgery
* need for a vessel sealing device during surgery

Exclusion Criteria:

* non able to understand informed consent or missing consent
* age <18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for laparoscopic visceral or gynecologic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Intra- and postoperative device-related complications | 30 days
Use of additional vessel sealing devices | one day

SECONDARY OUTCOMES:
Perioperative Blood Loss | 30 days
Duration of Surgery | one day

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Baselland Bruderholz, Bruderholz, Switzerland